CLINICAL TRIAL: NCT06417671
Title: The Effect of Postbiotics Supplementation on Exercise-induced Oxidative Stress.
Acronym: PB-EIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: PostBiotics-Exercise
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Postbiotics Supplement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization of the participants to the supplement or placebo condition will be performed via a random integer set generator (Random.org) available online.
  Neither the participants, nor the supplement provider will be aware of whether participants receive the postbiotic supplement or the placebo. Additionally, blood samples will be masked during the biochemical analysis, and during the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postbiotics supplementation (Experimental): Supplementation of postbiotics for 4 weeks
  Interventions: Dietary Supplement: Postbiotics supplementation
- Placebo supplementation (Placebo Comparator): Supplementation of placebo for 4 weeks
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Postbiotics supplementation — The participants will consume one capsule per day.
  Arms: Postbiotics supplementation
Dietary Supplement: Placebo supplementation — The participants will consume one capsule per day.
  Arms: Placebo supplementation

SUMMARY:
Scientific data on the effect of supplementation of postbiotics on exercise-induced oxidative stress are scarce. The main purpose of the research is to investigate the effect of postbiotics supplementation on exercise-induced oxidative stress and performance indicators after intense exercise. The study will be a cross-over, randomized, double-blind, controlled study that will be conducted in two cycles. Participants will be randomly assigned into one of the two trials: i) Postbiotics supplementation for 4 weeks, ii) Placebo supplementation for 4 weeks. Participants will then perform a 45-min treadmill running at (-15% slope, ~70% VO2max) followed by a time-trial (0% slope, ~95% VO2max) until exhaustion. Before, as well as 24 h, 48 h and 72 h after the exercise, participants will undergo measurements of exercise-induced muscle damage (EIMD) [delayed onset of muscle soreness (DOMS), creatine kinase], blood redox status [total antioxidant capacity, catalase, protein carbonyls, reduced glutathione, oxidized glutathione], and isokinetic performance (knee-extensors and knee-flexors isometric, concentric, eccentric torque) evaluation. In addition, metabolism (lactic acid) will be assessed before and 4 min after exercise. Afterwards, the participants will receive the postbiotics supplement or the placebo for 4 weeks, and will repeat the exercise protocol and measurements of EIMD, blood redox status and performance indices at the same time-points. At the second cycle, the participants will repeat the above procedures under the remaining condition. Between conditions, there will be a 14-day washout period. The results of the research will provide important information for coaches and physically active individuals, regarding the effectiveness of postbiotics in alleviating oxidative stress and improving performance after intense exercise.

DETAILED DESCRIPTION:
Acute, vigorous and/or unaccustomed exercise can induce muscle injury and oxidative stress. At moderate concentrations, reactive oxygen and nitrogen species (RONS) act as signaling molecules and promote adaptations to systematic training. Conversely, excessive production of RONS may cause destructive effects, due to the oxidation of important biomolecules such as lipids and proteins, but also DNA. Disruption of the redox balance can bring about adverse effects on exercise-induced adaptations, such as muscle damage and fatigue. For this reason, many professional as well as amateur athletes, often consume nutritional supplements such as antioxidants, anticipating to reduce inflammation and oxidative stress after intense exercise.

The human gastrointestinal tract is inhabited by various microorganisms, called the gut microbiome (GM). GM, among other things, contributes to the normal functioning of the immune system, contributes to the production of short-chain fatty acids (SCFAs) and vitamin synthesis as well as the digestion and absorption of food, protects against enteropathogens and regulates inflammatory and redox responses. Recent evidence also suggests that GM may be involved in athletic performance. In contrast, disruption of GM composition (dysbiosis) is characterized by reduced diversity, reduced abundance of health-promoting bacteria, and increased abundance of gram-negative and other pathogenic bacteria and is associated with various metabolic diseases such as obesity, diabetes, and various forms of cancer, systemic inflammation, oxidative stress and reduced performance. Thus, the supplementation of several "biotics" has been emerged as a means to regulate the GM in favor of health-promoting bacteria.

Postbiotics is defined as a "preparation of inanimate microorganisms and/or their components that confers a health benefit on the host". Evidence suggests that supplementation with postbiotics may regulate the GM, and consequently, strengthen the immune system, reduce intestinal permeability, improve antioxidant mechanisms, as well as accelerate recovery after exercise-induced inflammation, enhance adaptations to exercise, and improve performance. However, the scientific data regarding the possible beneficial effect of supplemental administration of postbiotics is limited. More research is needed, in order to determine the role of postbiotics supplementation on exercise-induced inflammation and redox status, but also on performance after intense exercise.

This study will investigate the potential of postbiotics supplementation to affect the recovery of exercise-induced oxidative stress and performance following intense, eccentrically biased acute exercise.

The study will be cross-over, randomized, double-blind, controlled, and will be conducted in two cycles. The participants, will be primarily informed of the study procedures, as well as the benefits and possible risks, they will also sign an informed consent form for participation in the study. Before the experimental procedure, they will be involved in a week of familiarization to the evaluation tests and the exercise protocol, at a low intensity. In addition, the participants will record their diet via a 7-days recall before their participation in the first experimental condition, and dietary data will be analyzed with ScienceFit Diet 200A diet analysis program (Science Technologies, Athens, Greece), in order to estimate that they do not consume nutrients that may affect muscle injury, inflammation and oxidative stress (e.g. antioxidants, etc.). Baseline measurements will take place at the Laboratory of Biochemistry, Physiology and Nutrition of Exercise (SmArT Lab), Department of Physical Education and Sports, University of Thessaly: anthropometric characteristics (body height, body mass, body mass index) via a stadiometer-scale (Stadiometer 208; Seca, Birmingham, UK), body composition (amount of body fat, lean body mass, fat mass, bone density) via by dual emission X-ray absorptiometry (DXA, GE-Healthcare, Lunar DPX NT, Belgium), aerobic capacity (VO2max) via an automated online pulmonary gas analyzer (Vmax Encore 29, BEBJO296, Yorba Linda, CA, USA) during a graded exercise protocol on a treadmill (Stex 8025T, Korea), isokinetic strength (isometric, concentric and eccentric torque of the knee extensors and knee flexors) on an isokinetic dynamometer (Cybex, HUMAC NORM 360, Ronkonkoma, NY), and muscle power via the assessment of countermovement jump (CMJ) via an optical measurement system (Optojump next, Microgate, USA). Participants will then be randomized in one of the two conditions: i) Postbiotics supplementation (50mg/day of Heat-killed Lactobacillus plantarum L-137, Immuno-LP20TM) for 4 weeks, or ii) placebo supplementation for 4 weeks. Randomization of the conditions will be done by a software generating random integers available on the internet (Random.org). Seven days later, participants will perform an exercise protocol comprised of 45 min downhill running (-15% slope, ~70-75% VO2max) on a treadmill followed by a time-trial (0% slope, ~95% VO2max) until exhaustion. Before the exercise protocol, as well as 24 h, 48 h and 72 h after exercise, delayed onset of muscle soreness (DOMS) via palpation of the knee extensors and knee flexors on a scale of 1 to 10 (1 = no pain at all; 10 = extreme pain), and muscle performance (CMJ, isometric, concentric and eccentric torque of the knee extensors and knee flexors) will be assessed. Additionally, blood samples will be collected at the same time-points for the assessment of creatine kinase (CK), and blood redox status [reduced glutathione (GSH), oxidized glutathione (GSSG), GSH/GSSG ratio, total antioxidant capacity (TAC), catalase (CAT), protein carbonyls (PC), uric acid, bilirubin)]. Furthermore, metabolism (lactic acid) will be assessed before and 4 min after exercise by analyzing capillary blood with a portable lactate analyzer (Lactate Plus, Nova Biomedical, USA). After a 14-days washout period, participants will repeat the exact same procedures for the remaining condition in the second cycle. Additionally, the 7-day diet recall will be given to the participants to follow the same diet before the experimental exercise protocol at the second cycle.

ELIGIBILITY:
Inclusion Criteria:

* Physically active subjects (VO2max ≥35ml/kg/min)
* Absence of musculoskeletal injury (≥6 months)
* Abstinence from the use of ergogenic supplements (≥1 month)
* Abstinence from anti-inflammatory drugs (≥1 month)
* Abstinence from pre-pro-postbiotic supplements (≥6 months)
* Abstinence from participating in exercise with eccentric content for at least 7 days before exercise
* Abstinence from alcohol and energy drinks before exercise

Exclusion Criteria:

* Recent history of musculoskeletal injury (<6 months)
* Use of ergogenic performance supplements (<1 month)
* Taking anti-inflammatory drugs (<1 month)
* Taking pre-pro-postbiotic supplements (<6 months)
* Participation in exercise with eccentric content in the previous 7 days before exercise
* Consumption of alcohol and energy drinks before exercise

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in PC | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of PC will be measured in plasma
Changes in malondialdehyde (MDA) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of MDA will be measured in plasma
Changes in reduced glutathione (GSH) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of GSH will be measured in red blood cells
Changes in oxidized glutathione (GSSG) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of GSSG will be measured in red blood cells
Changes in GSH/GSSG ratio | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  GSH/GSSG ratio will be calculated
Changes in catalase | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of catalase will be measured in red blood cells
Changes in total antioxidant capacity (TAC) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  TAC will be measured in plasma
Changes in uric acid | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of uric acid will be measured in plasma
Changes in bilirubin | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Concentration of bilirubin will be measured in plasma
Changes in blood lactate | At baseline (pre), and 4 min post-trial
  Concentration of lactate will be measured in capillary blood
Changes in in delayed onset of muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Muscle soreness of the KF and KE will be assessed via palpation of the muscle belly and the distal regions following 3 squats, and the subjective pain will be recorded on a 10-point scale (1 = no pain, 10 = extreme pain)
Changes in creatine kinase (CK) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  CK will be will be measured in serum
Changes in countermovement jump (CMJ) height | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  CMJ height will be measured with an optical system
Changes in isokinetic strength of knee extensors (KE) and knee flexors (KF) | At baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-exercise
  Isometric, concentric and eccentric peak torque of the KE and KF of both limbs will be assessed on an isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Principal Investigator — University of Thessaly, DPESS
Locations (1):
- Department of Physical Education and Sport Science, Uninersity of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jamurtas AZ, Garyfallopoulou A, Theodorou AA, Zalavras A, Paschalis V, Deli CK, Nikolaidis MG, Fatouros IG, Koutedakis Y. A single bout of downhill running transiently increases HOMA-IR without altering adipokine response in healthy adult women. Eur J Appl Physiol. 2013 Dec;113(12):2925-32. doi: 10.1007/s00421-013-2717-5. Epub 2013 Sep 26. PMID 24068487
- [Result] Deli CK, Fatouros IG, Paschalis V, Tsiokanos A, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. Iron Supplementation Effects on Redox Status following Aseptic Skeletal Muscle Trauma in Adults and Children. Oxid Med Cell Longev. 2017;2017:4120421. doi: 10.1155/2017/4120421. Epub 2017 Jan 22. PMID 28203319
- [Result] Deli CK, Poulios A, Georgakouli K, Papanikolaou K, Papoutsis A, Selemekou M, Karathanos VT, Draganidis D, Tsiokanos A, Koutedakis Y, Fatouros IG, Jamurtas AZ. The effect of pre-exercise ingestion of corinthian currant on endurance performance and blood redox status. J Sports Sci. 2018 Oct;36(19):2172-2180. doi: 10.1080/02640414.2018.1442781. Epub 2018 Feb 22. PMID 29469654
- [Result] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Result] Sales KM, Reimer RA. Unlocking a novel determinant of athletic performance: The role of the gut microbiota, short-chain fatty acids, and "biotics" in exercise. J Sport Health Sci. 2023 Jan;12(1):36-44. doi: 10.1016/j.jshs.2022.09.002. Epub 2022 Sep 9. PMID 36089243
- [Result] Jager R, Mohr AE, Carpenter KC, Kerksick CM, Purpura M, Moussa A, Townsend JR, Lamprecht M, West NP, Black K, Gleeson M, Pyne DB, Wells SD, Arent SM, Smith-Ryan AE, Kreider RB, Campbell BI, Bannock L, Scheiman J, Wissent CJ, Pane M, Kalman DS, Pugh JN, Ter Haar JA, Antonio J. International Society of Sports Nutrition Position Stand: Probiotics. J Int Soc Sports Nutr. 2019 Dec 21;16(1):62. doi: 10.1186/s12970-019-0329-0. PMID 31864419
- [Result] Salminen S, Collado MC, Endo A, Hill C, Lebeer S, Quigley EMM, Sanders ME, Shamir R, Swann JR, Szajewska H, Vinderola G. The International Scientific Association of Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of postbiotics. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):649-667. doi: 10.1038/s41575-021-00440-6. Epub 2021 May 4. PMID 33948025
- [Result] Lee CC, Liao YC, Lee MC, Cheng YC, Chiou SY, Lin JS, Huang CC, Watanabe K. Different Impacts of Heat-Killed and Viable Lactiplantibacillus plantarum TWK10 on Exercise Performance, Fatigue, Body Composition, and Gut Microbiota in Humans. Microorganisms. 2022 Nov 3;10(11):2181. doi: 10.3390/microorganisms10112181. PMID 36363775